CLINICAL TRIAL: NCT01537146
Title: Examination of the LIA (Local Infiltration) Versus Regional Blockade as Pain Management for Open-wedge High Tibial Osteotomy
Brief Title: Local Infiltration Versus Block Against Pains After High Tibial Osteotomy
Acronym: HTO_pains
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ON-04-019-ACL
Record Dates: First submitted 2011-08-02; First posted 2012-02-23 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis; Malalignment
Keywords: unicompartmental; osteoarthritis; varus; malalignment; opening wedge; HTO; high; tibia; osteotomy
MeSH Terms: conditions — Osteoarthritis | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral Block (Active Comparator)
  Interventions: Drug: Ropivacaine
- Local Infiltration Anagesia (Active Comparator)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Bolus infusion via catheter/6H for 24H
  Other Names: No other names
  Arms: Femoral Block
Drug: Ropivacaine — Intra operational bolus infusion. Bolus infusion via catheter /6H for 24H
  Other Names: no other names
  Arms: Local Infiltration Anagesia

SUMMARY:
The purpose of this study is to elucidate whether patients operated with high tibia open-wedge osteotomy for osteoarthritis of the knee can be treated more appropriately, so that both healing and rehabilitation are served optimally.

DETAILED DESCRIPTION:
Axis corrective surgery of the knee is an attractive alternative to the knee prosthesis in young active patients with unilateral osteoarthritis of the knee. The purpose of this study is to elucidate whether patients operated with high tibia open-wedge osteotomy for osteoarthritis of the knee pain can be treated more appropriately, so that both healing and rehabilitation are served optimally.

Proximal open-wedge tibia osteotomy is an accepted treatment option for younger patients with unilateral osteoarthritis of knee. 70 such operations are performed in the investigators Orthopaedic Divisions each year. The surgery involves cutting through the upper end of the tibia and opens the bone using specialized instruments. The tibia is lengthened on the medial side with the purpose of correcting the mechanical axis of the knee joint. The surgery is associated with many pains in the early postoperative phase. Until now, pain treatment has been controlled with either epidural block, or regional block via femoral catheter. Both treatments may involve risks such as loss of strength and sensibility disturbance, which often prolongs the early recovery and mobilization. Moreover, pain treatment administered via femoral catheter is often not sufficient as a part of the area behind the knee joint is not covered.

With the advent of new pain therapies, particularly intra operative administration of local anaesthetics directly in the operating field and catheter administration for postoperative pain management, there is hope that those disadvantages are eliminated. By ensuring an effective pain treatment and the possibility of early mobilization only hours after completion of surgery, this will allow for better patient care in terms of reduced pain, shorter hospitalization and quicker rehabilitation.

New results show that the healing of bone opening is not compromised by rapid mobilization. The migration of bone parts around the opening is measured by roentgen stereometric analysis (RSA), with a precision of approximately 0.2 mm. This verifies stable healing of the bone opening.

ELIGIBILITY:
Inclusion Criteria:

* Planned primary open-wedge high tibia osteotomy
* Patients (male/female) ≥ 18 år
* Patients giving written informed consent and authority.
* Patients receiving epidural anaesthesia

Exclusion Criteria:

* Patients with intolerance to trial medications
* Rejection of or contraindicated epidural anaesthesia
* Patients with rheumatoid arthritis.
* Patients with Body Mass Index (BMI) ≥ 35
* Patients that do not read or write Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PN morphine consumption | Hours (up to 24 hours)
  Use of morphine recorded in medicine journal

SECONDARY OUTCOMES:
Pain | Hours (up to 24 hours)
  Level of pain experienced by the patient, recorded by NRS (numerical rank scale)
Knee Function | Months (up to 16 months)
  Knee function in the patient, measured by KOOS questionnaire
General Health Parameters | Months (up to 16 months)
  General Health Parameters, measured by EQ-5D questionnaire
Stability in the osteotomy | Months (up to 16 months)
  Stability in the opening-wedge osteotomy, measured with RSA (Rontgen Stereometric Analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Anders C Laursen, MD, Principal Investigator — Northern Orthopaedic Division, Denmark; Mogens B Laursen, MD, PhD, Study Chair — Northern Orthopaedic Division, Denmark
Locations (1):
- Northern Orthopaedic Division, Clinik Farsoe, Aalborg University Hospital, Farsø, Northern Jutland, Denmark